CLINICAL TRIAL: NCT05238428
Title: Mind the Vaccination Gap: Understanding and Overcoming the Racial/Ethnic Inequalities in COVID-19 Vaccination Acceptance
Brief Title: Understanding and Overcoming the Racial/Ethnic Inequalities in COVID-19 Vaccination Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Essex (Other)
Collaborators: University of Southern California (Other); Department of Health and Social Care (Unknown); Kingston University (Other)
Responsible Party: Principal Investigator, Marie Juanchich, Reader/Associate Professor in Psychology, University of Essex
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETH2122-0265
Record Dates: First submitted 2022-02-01; First posted 2022-02-14 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Vaccine Refusal
Keywords: COVID-19 vaccination acceptance; vaccine hesitancy; trust; health inequality; racial/ethnicity
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: In a 4 x 4 experimental design, the investigators will manipulate the content of the vaccination invitation message in within-subject and the message source in between-subjects. Each participant will hence read four versions of the COVID-19 booster vaccination invitation message sent by one of the four possible sources.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will read and evaluate 4 versions of the vaccination invitation. The condition will be selected randomly by the Qualtrics algorithm (with an even selection rate). The four invitations will be presented to each participant in a random order based on the Qualtrics randomisation algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Control sender + control content (No Intervention): Participants will read the following text in an online survey:
  You are invited to book your COVID-19 booster vaccination. Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
- Control sender + Low trust boost content (Experimental): Participants will read the following text in an online survey:
  You are invited to book your COVID-19 booster vaccination. The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Control sender + Medium trust boost content (Experimental): Participants will read the following text in an online survey:
  You are invited to book your COVID-19 booster vaccination. The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  Vaccines may cause side effects, but the benefits outweigh the risks. The most common side effects are very mild (e.g., sore arm, fever) and severe side effects are very rare (e.g., allergic reaction).
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Control sender+ high trust boost content (Experimental): Participants will read the following text in an online survey:
  You are invited to book your COVID-19 booster vaccination. The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  This vaccination is especially important for people who are at higher risk from COVID such as older individuals or those from ethnic minorities.
  Vaccines may cause side effects, but the benefits outweigh the risks. The most common side effects are very mild (e.g., sore arm, a fever) and severe side effects are very rare (e.g., allergic reaction).
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Low trust boost Sender + control content (Experimental): Participants will read the following text in an online survey:
  As your local GP, I would like to invite you to book your COVID-19 booster vaccination.
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Low trust boost Sender + low trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Low trust boost Sender + medium trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  Vaccines may cause side effects, but the benefits outweigh the risks. The most common side effects are very mild (e.g., sore arm, fever) and severe side effects are very rare (e.g., allergic reaction).
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Low trust boost sender + high trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  This vaccination is especially important for people who are at higher risk from COVID such as older individuals or those from ethnic minorities.
  Vaccines may cause side effects, but the benefits outweigh the risks. The most common side effects are very mild (e.g., sore arm, a fever) and severe side effects are very rare (e.g., allergic reaction).
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Medium trust boost Sender + control content (Experimental): Participants will read the following text in an online survey:
  As your local GP and a health expert who cares for the local community, I would like to invite you to book your COVID-19 booster vaccination.
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Medium trust boost sender + low trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP and a health expert who cares for the local community, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Medium trust boost sender + Medium trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP and a health expert who cares for the local community, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  Vaccines may cause side effects, but the benefits outweigh the risks. The most common side effects are very mild (e.g., sore arm, fever) and severe side effects are very rare (e.g., allergic reaction).
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- Medium trust boost Sender+ high trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP and a health expert who cares for the local community, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  This vaccination is especially important for people who are at higher risk from COVID such as older individuals or those from ethnic minorities.
  Vaccines may cause side effects, but the benefits outweigh the risks. The most common side effects are very mild (e.g., sore arm, a fever) and severe side effects are very rare (e.g., allergic reaction).
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Interventions: Behavioral: Trust boost
- High trust boost sender + control content (Experimental): Participants will read the following text in an online survey:
  As your local GP and a health expert who cares for the local community, I would like to invite you to book your COVID-19 booster vaccination.
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Dr Sanjay Kumar
  Interventions: Behavioral: Trust boost
- High trust boost sender + low trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP and a health expert who cares for the local community, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Dr Sanjay Kumar
  Interventions: Behavioral: Trust boost
- High trust boost Sender + medium trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP and a health expert who cares for the local community, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  Vaccines may cause side effects, but the benefits outweigh the risks. The most common side effects are very mild (e.g., sore arm, fever) and severe side effects are very rare (e.g., allergic reaction).
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Dr Sanjay Kumar
  Interventions: Behavioral: Trust boost
- High trust boost sender + high trust boost content (Experimental): Participants will read the following text in an online survey:
  As your local GP and a health expert who cares for the local community, I would like to invite you to book your COVID-19 booster vaccination.
  The vaccine reduces your chance of becoming infected and protects you against severe forms of the illness. It also protects your loved ones by reducing the risk that you infect others. COVID can be severe, don't risk it.
  This vaccination is especially important for people who are at higher risk from COVID such as older individuals or those from ethnic minorities.
  Vaccines may cause side effects, but the benefits outweigh the risks. The most common side effects are very mild (e.g., sore arm, a fever) and severe side effects are very rare (e.g., allergic reaction).
  Click here to book an appointment: accurx.thirdparty.nhs.uk/r/aafwaczmd5
  Dr Sanjay Kumar
  Interventions: Behavioral: Trust boost

INTERVENTIONS:
Behavioral: Trust boost — The investigators adapt the wording of the vaccination invitation to foster trust and increase vaccination acceptance.
  Arms: Control sender + Low trust boost content; Control sender + Medium trust boost content; Control sender+ high trust boost content; High trust boost Sender + medium trust boost content; High trust boost sender + control content; High trust boost sender + high trust boost content; High trust boost sender + low trust boost content; Low trust boost Sender + control content; Low trust boost Sender + low trust boost content; Low trust boost Sender + medium trust boost content; Low trust boost sender + high trust boost content; Medium trust boost Sender + control content; Medium trust boost Sender+ high trust boost content; Medium trust boost sender + Medium trust boost content; Medium trust boost sender + low trust boost content

SUMMARY:
With the constant threat of new epidemic waves and the emergence of variants, COVID-19 resilience can only be attained when a sufficient level of immunity is achieved. Yet, in the US and the UK, COVID-19 vaccination campaigns have failed to secure consistent vaccination acceptance in racial/ethnic minority communities. Despite racial/ethnic minorities being more at risk from COVID-19, they are less vaccinated than the White majority. The investigators propose that current vaccination invitation messages are deemed less trustworthy by racial/ethnic minorities than the White majority and that this might partly explain reduced vaccination acceptance. To provide causal evidence of the role of trust and actionable insights, the investigators will experimentally assess the benefits of new invitation messages to receive the COVID-19 booster dose in large, racially/ethnically diverse samples in the US and the UK. Results will evidence how to increase message and source trustworthiness to foster trust and vaccination acceptance across racial/ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* if participants complete the study in less than 5 minutes
* if participants complete the study without paying attention (as indicated by their answers to two attention check questions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4039 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Trust perception | immediately after intervention
  Perceived trustworthiness of the vaccine invitation. Participants will rate how trustworthy is the invitation message on a 5 point Likert scale (1: Untrustworthy 3: Not sure, 5: Trustworthy)
Vaccination appointment booking | immediately after intervention
  Likelihood to book a vaccination appointment via the message. Participants will report if they would use the link in the message to book their vaccination appointment on a 5 point Likert scale (1: No, I would not, 3: Not sure/maybe later, 5: Yes, I would)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Juanchich, PhD, Study Chair — University of Essex
Locations (1):
- Qualtrics. The data is gathered via an online platform., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data of the study will be shared on the Open Science Framework after publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data and the study protocol will be shared after the main scientific output is accepted (possibly pending revision). The investigators anticipate this would be early 2023.
Access Criteria: The data and study protocol will be free to access to the public